CLINICAL TRIAL: NCT07296718
Title: Evaluation of the Clinical and Growth-related Effects of Probiotics in Preterm Infants: A Randomized, Placebo Controlled Clinical Trial.
Brief Title: Single Vs Multi-strain Probiotics for Preterm Neonates
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Madiha, MPhil (Other)
Responsible Party: Sponsor-Investigator, Madiha, MPhil, Co-investigator, The Islamia University of Bahawalpur, Khawaja Fareed CampusDr
Organization: The Islamia University of Bahawalpur, Khawaja Fareed CampusDr (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: NEOPRO-SvsM
Record Dates: First submitted 2025-11-19; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Necrotizing Enterocolitis of Newborn; Sepsis Newborn; Growth; Feeding Intolerance
Keywords: Probiotics; Preterm neonates; Single vs Multiple strain
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Intervention Model Description: Placebo-controlled randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- P1 (Placebo Comparator): 1 ml of 10% dextrose water will be dispensed in 5cc syringe and administered orally or via feeding tube for 28 days.
  Interventions: Dietary Supplement: Dextrose 10%
- P2 (Active Comparator): Single strain probiotic- Lactobacillus rhamnosus GG. The single dose 1.5×109 CFU/day as 1 mL of the reconstituted solution will be given every day via the feeding tube or orally as applicable until reaching feeds of 50 mL/kg/day. It will be increased thereafter to 3×109 CFU/day once feeds exceed 50mL/kg/day.
  Interventions: Drug: Lactobacillus Rhamnosus GG
- P3 (Active Comparator): Multiple strain probiotic-Bifidobacterium BB-12, Lactobacillus paracasei, L casei-431, Streptococcus thermophilus TH-4.
  The single dose 1.5×109 CFU/day as 1 mL of the reconstituted solution will be given every day via the feeding tube or orally as applicable until reaching feeds of 50 mL/kg/day. It will be increased thereafter to 3×109 CFU/day once feeds exceed 50mL/kg/day.
  Interventions: Drug: Bifidobacterium BB-12, Lactobacillus paracasei, L casei-431, Streptococcus thermophilus TH-4

INTERVENTIONS:
Dietary Supplement: Dextrose 10% — P1
  Other Names: Placebo
  Arms: P1
Drug: Lactobacillus Rhamnosus GG — Single Strain
  Other Names: Prepro GG
  Arms: P2
Drug: Bifidobacterium BB-12, Lactobacillus paracasei, L casei-431, Streptococcus thermophilus TH-4 — Multiple Strain
  Other Names: Amybact
  Arms: P3

SUMMARY:
The goal of this randomized control clinical trial is to determine if probiotics can prevent mortality and morbidity in preterm neonates. It also evaluates effects of probiotics on feeding pattern and growth. It will also learn about the comparative effects of single vs multiple strain probiotics.

It aims to answer:

Does probiotics improve the health and growth outcomes in preterm neonates in our population? Does single vs multiple strain of probiotics have difference in effects?

Participants will:

Participants given either single strain or multiple strain probiotics for 28 days post birth.

Data about mortality, morbidity, feeding pattern and growth (weight, height, head circumference gain) recorded on daily basis.

DETAILED DESCRIPTION:
This trial is single-centered, parallel, multi-arm, 1:1:1 randomized, blinded, placebo controlled clinical trial. It compares 3 groups; Group P1 (Placebo), Group P2-Single Strain probiotic (Lactobacillus rhamnosus GG) and Group P3- Multiple strains probiotic ( Bifidobacterium BB-12, Lactobacillus paracasei, L casei-431, Streptococcus thermophilus TH-4) for preventing preterm neonatal morbidities, improving feeding tolerance and overall growth.

Primary objective: The primary objective of our trial will be to compare the incidence and severity of Necrotizing enterocolitis (NEC) from the time of trial participation till the end of trial treatment (28 days) according to Bell's grading criteria.

Secondary objectives:

All these outcomes will be measured from the day intervention started to the end of supplementation (28 days)

* To evaluate incidence of sepsis, intracerebral haemorrhage and periventricular leukomalacia, retinopathy of prematurity and bronchopulmonary dysplasia)
* To estimate the time to full enteral feeding (i.e., ≥150 ml/kg/day) and feeding tolerance based on Davy's Neonatal Feeding Assessment Scale (NFAS).
* To determine the effect of probiotics on growth (weight, height, and head circumference) of premature babies
* To assess comparative efficacy of single strain vs combination probiotics for aforementioned objectives

Framework/hypothesis: The experimental group P2 (Lactobacillus rhamnosus GG) and Group P3- ( Bifidobacterium BB-12, Lactobacillus paracasei, L casei-431, Streptococcus thermophilus TH-4) are superior to control group (Placebo) as preventing NEC and other morbidities in preterm neonates, thus improving feeding tolerance and overall growth.

ELIGIBILITY:
Inclusion Criteria:

Preterm babies of gestational age <35+6days, birth weight <2500 grams, received and tolerated at-least one feed within 72 hours of birth and informed consent from parents or guardian.

Exclusion Criteria:

* Neonates with major congenital malformations, gastrointestinal anomalies, early onset sepsis (C-reactive protein (CRP) >10 mg/L in the first 72 h of life) and renal insufficiency

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 249 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Necrotizing enterocolitis (NEC) | From the day intervention started to day 28 of supplementation
  Bell's classification used for grading and diagnosis

SECONDARY OUTCOMES:
Neonatal Sepsis | From the day intervention started to day 28 of supplementation
  Clinical sepsis is defined as condition with at least two signs of systemic inflammatory response (e.g. temperature >38 C or <36.5 C, tachycardia > 200/min etc.), one laboratory sign (e.g. C-reactive protein >20mg/L) but no proof of causative agent in blood culture. Clinical sepsis with proof of blood culture positive for causative agent was defined as confirmed sepsis.
Feeding Intolerance | From the day intervention started to day 28 of supplementation
  A gastrointestinal tolerance score, based on gastric residual volume, emesis, abdominal distension, number of stools and nil per oral days was calculated to identify and score feeding intolerance. Each score as 1. A score of >2 was considered gastric intolerance.
Weight | From the day intervention started to day 28 of supplementation
  Weight measured in grams
Body length | From the day intervention started to day 28 of supplementation
  Measured in millimeters daily once
Head Circumference | From the day study started to day 28 of supplementation
  Measured in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Imran Masood, PhD, Principal Investigator — The Islamia University of Bahawalpur, Khawaja Fareed Campus
Locations (1):
- Bahawal Victoria Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT07296718/ICF_000.pdf